CLINICAL TRIAL: NCT01142310
Title: Reversing Corticosteroid Induced Memory Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sherwood Brown, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 122009-028; R01MH082845 (NIH)
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Memory Impairment
MeSH Terms: conditions — Memory Disorders | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamotrigine (Active Comparator): Dose titration: begin at Baseline at 25mg PO QD for two weeks. Increase to 50mg PO QD at Week 2 for two weeks. Increase to 100mg PO QD at Week 4. Increase to 150mg PO QD at Week 5. Increase to 200mg PO QD at Week 6. Increase to 250mg PO QD at Week 7. Increase to 300mg PO QD at Week 8. Increase to 350mg PO QD at Week 9. Increase to 400mg PO QD at Week 10. Stay at 400mg PO QD from Week 10 to Week 48.
  Interventions: Drug: Lamotrigine
- Placebo (Placebo Comparator): Placebo administered the same as the Lamotrigine just described.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine will be initiated at 25 mg/day and upwardly titrated to a dose of 400 mg/day over 10 weeks.
  Other Names: Lamictal
  Arms: Lamotrigine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Medically stable outpatients receiving chronic oral corticosteroid therapy were enrolled in a 48-week randomized, double-blind, placebo-controlled, parallel-group, trial of lamotrigine.

DETAILED DESCRIPTION:
Stress and corticosteroid exposure are associated with changes in both the human and animal hippocampus. An extensive literature suggests that corticosteroid-induced changes in the hippocampus are, in part, mediated through increases in extracellular glutamate. In animals, agents that decrease glutamate release prevent dendritic changes in the hippocampus secondary to stress or corticosterone. We have developed a research program using patients receiving prescription corticosteroids (e.g., prednisone) to explore the effects of corticosteroids on the human hippocampus. Our research program is translational in focus, with a goal of exploring whether the reported effects of corticosteroids on the animal hippocampus are also found in humans. A current focus of our research is examining glutamate release inhibitors in patients taking corticosteroids. We have both open-label and placebo-controlled pilot data suggesting that the glutamate release inhibitor lamotrigine is associated with significant improvement in declarative memory (a measure of hippocampal performance) in this population. A definitive study examining declarative memory in corticosteroid-dependent patients receiving lamotrigine vs. placebo is proposed. Neuroimaging and mood will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* English-speaking men and women
* Physician diagnosis of any chronic medical condition requiring treatment with oral corticosteroids confirmed by chart review and/or patients assessment by the PI or co-I.s.
* Receiving prednisone therapy of at least 5 mg of prednisone daily for at least 6 months with anticipated treatment for ≥ 15 additional months.

Exclusion Criteria:

* Baseline RAVLT total T-Score ≥ 60
* Illnesses associated with CNS involvement (e.g., multiple sclerosis, lupus, seizures, brain tumors, head injury with loss of consciousness of more than 30 minutes) or cognitive impairment (e.g., lifetime drug or alcohol dependence, schizophrenia, and mood disorders - e.g., bipolar disorder, major depressive disorder) that appear to be unrelated to corticosteroid use or history of ventilator use that suggests hypoxia. We will include patients with lupus if they do not appear, based on medical history and discussion with treating physician, have significant CNS involvement. We will include participants with brief loss of consciousness. In prior studies we have found that many otherwise eligible participants were excluded due to very brief LOC in childhood or in a motor vehicle accident.
* Mental retardation or other severe cognitive impairment.
* Pregnant or nursing women.
* Severe or life-threatening medical illness that would make completion of study unlikely or study participation potentially unsafe (e.g., highly unstable asthma requiring frequent hospitalization)
* Contraindications to lamotrigine therapy (severe side effects in the past, taking medications such as some anticonvulsants with drug-drug interactions with lamotrigine).
* High risk or danger to self or others as defined by > 1 lifetime suicide attempt or assault, any suicide attempt or assault within the past year, and active suicidal or homicidal ideation that includes a plan and intent
* Therapy with medications (valproate, carbamazepine, primidone, phenytoin, rifampin, phenobarbital) that alter the metabolism of lamotrigine
* Metal implants, claustrophobia, or other contraindications to MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System (Asthma, Allergy, & Arthritis Clinics), Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine: Participants took 25mg of Lamotrigine PO QD for two weeks. Dose was increased to 50mg PO QD at Week 2 for two weeks. Increased to 100mg PO QD at Week 4. Increased to 150mg PO QD at Week 5. Increased to 200mg PO QD at Week 6. Increased to 250mg PO QD at Week 7. Increased to 300mg PO QD at Week 8. Increased to 350mg PO QD at Week 9. Increased to 400mg PO QD at Week 10. Participants stayed at 400mg PO QD from Week 10 to Week 48.
- Placebo: Placebo was administered the same as the Lamotrigine dose titration described.
Period: Overall Study
Arm/Group | Lamotrigine | Placebo
Started | 26 | 28
Completed | 17 | 16
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine: Participants took Lamotrigine beginning at 25mg/day and increased to a dose of 400mg/day over 10 weeks using a fixed scheduled.
- Placebo: Placebo administered the same as the Lamotrigine.
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.192 (11.771) | 46.286 (9.974) | 44.315 (10.968)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 15 | 28
  White | 13 | 12 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Rey Auditory Verbal Learning Test (RAVLT)
Description: The Rey Auditory Verbal Learning Test (RAVLT) measures verbal or declarative learning and memory. The test consists of 15 nouns read aloud for five consecutive trials with each trial followed by a free-recall trial. Following the fifth trial, an interference list of 15 different words is presented followed by a free-recall trial of that list. Delayed recall of the first list is tested immediately following the interference list and after a 20-minute delay. A recognition test of 50 words including the 15 original words is presented after the delayed recall. Equivalent, alternative versions (different words) were used to minimize practice or learning effects from repeated administration. The raw scores (number of words correct across trials 1-5) are converted to standardized T-scores (M=50; SD=10). This score is used to determine the participant's performance in relation to norm-referenced expectations based on age and sex. A higher score reflects better performance.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 26 | 28
T Score | 45.741 (9.63) | 43.286 (6.57)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study between baseline and end of study procedures, up to 48 weeks.
Description: Adverse events were assessed by a weekly questionnaire at each appointment or when contacted by phone for a brief follow-up.
Groups:
- Lamotrigine: Participants took Lamotrigine beginning at 25mg PO QD and increased to a dose of 400mg PO QD over 10 weeks using a fixed scheduled.
- Placebo: Placebo was administered the same as Lamotrigine.
Arm/Group | Lamotrigine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/28
Serious Adverse Events (participants affected / at risk) | 5/26 | 6/28
Other Adverse Events (participants affected / at risk) | 2/26 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=26) | Placebo (N=28)
Cancer (General disorders) | 1 (1) | 0 (0) — Serious, unexpected, not related to medication study
Foot Amputation (Surgical and medical procedures) | 0 (0) | 1 (1) — Serious, unexpected, not related to medication study
Kidney Stone (Infections and infestations) | 0 (0) | 1 (1) — Serious, unexpected, not related to medication study
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Serious, unexpected, not related to medication study
Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Serious, unexpected, not related to medication study
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Serious, unexpected, not related to medication study
Vaginal Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Serious, unexpected, not related to medication study
Hypotension (Vascular disorders) | 0 (0) | 1 (1) — Serious, unexpected, not related to medication study
Bacterial Vaginosis (Infections and infestations) | 0 (0) | 1 (1) — Serious, unexpected, not related to medication study
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Serious, unexpected, not related to medication study
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Serious, unexpected, not related to medication study
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) — Serious, unexpected, not related to medication study
Influenza (Infections and infestations) | 1 (1) | 0 (0) — Serious, unexpected, not related to medication study
Kidney Biopsy (Surgical and medical procedures) | 1 (1) | 0 (0) — Serious, unexpected, not related to medication study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=26) | Placebo (N=28)
Fall (Social circumstances) | 1 (2) | 1 (1) — Not serious, unexpected, not related to medication study
Dizziness (General disorders) | 2 (2) | 0 (0) — Not serious, unexpected, not related to medication study
Car Acciddent (Social circumstances) | 0 (0) | 1 (1) — Not serious, unexpected, not related to medication study
Nose Bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not serious, unexpected, not related to medication study
Keratoconus (Eye disorders) | 1 (1) | 0 (0) — Not serious, unexpected, not related to medication study
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Not serious, unexpected, not related to medication study
Hypertension (Vascular disorders) | 1 (1) | 0 (0) — Not serious, unexpected, not related to medication study
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — Not serious, unexpected, not related to medication study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No